CLINICAL TRIAL: NCT00995995
Title: Evaluation of the Duration of Oral Combination Therapy in Type 2 Diabetes, Prior to the Initiation of Insulin in the UK
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113030
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients
  Interventions: Drug: Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone — Rosiglitazone

SUMMARY:
Carry out the cost-effectiveness analysis of rosiglitazone on a population in line with the rosiglitazone license and using UK costs

ELIGIBILITY:
Inclusion Criteria:

* Rosiglitazone Type II Diabetes studies

Exclusion Criteria:

* Studies without the required outcome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults - obtainable from the literature
Sampling Method: Probability Sample
Enrollment: 7641 (Actual)
Dates: Start 2008-10; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness of rosiglitazone | From literature

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline